CLINICAL TRIAL: NCT02133326
Title: Assessment of Preemptive Analgesic Effect of Caldolor® vs. Ofirmev® on Third Molar Surgery: A Prospective, Randomized, Double-blinded Clinical Trial
Brief Title: Efficacy Study of IV Ibuprofen vs IV Acetaminophen Post Surgical Extraction
Acronym: Caldolor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tufts University School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Caldolor vs. Orfimev Clinical
Record Dates: First submitted 2013-09-17; First posted 2014-05-08 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-10

CONDITIONS: Impacted Wisdom Teeth
Keywords: Analgesia; Third Molar Extraction; Ibuprofen; Acetaminophen; Pain Medicine; Nonsteroidal; Anti-inflammatory
MeSH Terms: conditions — Agnosia | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caldolor (Experimental): 800 mg of Caldolor® will be infused at the rate of 5-7 minutes as per the manufacturer's guidelines or
  Interventions: Drug: Caldolor
- Ofirmev (Experimental): 1000 mg of Ofirmev® will be infused at the rate of 15 minutes as per the manufacturer's guidelines.
  Interventions: Drug: Ofirmev

INTERVENTIONS:
Drug: Caldolor — Subject will be given Caldolor by IV prior to surgery.
  Other Names: IV Ibuprofen
  Arms: Caldolor
Drug: Ofirmev — Subject will be given Ofirmev prior to surgery.
  Other Names: Acetaminophen
  Arms: Ofirmev

SUMMARY:
This study will compare how effective a single dose of an intravenous (IV) ibuprofen is when compared to single dose of IV acetaminophen in reducing pain. We will administer this study medication thirty minutes prior to removal of wisdom teeth. We want to see if administering these drugs prior to surgery may reduce post-operative pain.

Administration of nonsteroidal anti-inflammatory drug before the onset of inflammation during surgery will reduce postoperative pain following third molar extraction when compared to the acetaminophen group. Subjects receiving nonsteroidal anti-inflammatory drug will consume less opioid medications compared to those receiving preemptive acetaminophen.

DETAILED DESCRIPTION:
The surgical removal of third molars is a common surgical procedure performed in dentistry. Surgery to extract an impacted third molar can be due to various reasons such as infection, caries, pain, cyst or tumor formation, or to facilitate orthodontic treatment. Both clinicians and patients are concerned with the postoperative pain following surgery.

Rationale for model selection The oral surgery model is well-suited for the measurement of acute pain.The model has been shown to be sensitive to the effects of analgesic drugs and is useful for examining peripheral biochemical measures of drugs in vivo.This model is recommended by the US Food and Drug Administration because patients are usually healthy without complicating medical conditions and most patients have pain for a short, predictable period after surgery.

Rationale for drug selection Pain from the surgical incision and tissue manipulation associated with the surgical procedure is instigated immediately. This gives way to inflammatory pain that follows inflammatory cell recruitment to the injured area within the course of several hours. Inflammatory pain generally continues for several days, depending on the nature of the surgical procedure. As a consequence of tissue damage and release of neurogenic inflammatory mediators, there is activation of specific receptors and pathways that can contribute to central sensitization and development of hyperalgesia and persistent pain. While various pharmacological strategies, including the use of opioids, provide adequate attenuation of pain, their use is associated with undesirable side effects, drug interactions, pharmacokinetic variability, and often inadequate dosing, all of which can lead to ineffective analgesia and prolonged suffering. Opioids do not interrupt the inflammatory component of pain.

The study drug Caldolor® is an intravenous formulation of ibuprofen which was approved by the FDA in June 2009. Caldolor® is the first injectable product available in the United States for the treatment of pain and fever. This is the first study in dentistry evaluating the use of Caldolor® as a preemptive analgesia. Southworth et al and colleagues randomized 406 patients undergoing elective single-site orthopedic or abdominal surgery to 400 mg intravenous (IV) Caldolor, 800 mg IV Caldolor, or placebo. The results showed that patients in the 800 mg group had a 25.6% lower median morphine use (P = .026) over the first 24 hours of treatment than the placebo group. Patients in the 400 mg group did not have a lower use of morphine, but both the 400 and 800 mg groups reported less pain at rest and with movement than with placebo.

The comparator group Ofirmev® is intravenous acetaminophen and was recently approved by the FDA for the management of mild to moderate pain, the management of moderate to severe pain with adjunctive opioid analgesics, and the reduction of fever. In a study conducted for total abdominal hysterectomy, preemptive IV paracetamol (acetaminophen) 1 g provided good quality postoperative analgesia, with decreased consumption of morphine and minimal side effects. Studies have showed that the use of 1 g of paracetamol as a single intravenous preemptive dose in abdominal surgery with perioperative epidural analgesia did not reduce the analgesic consumption and the intensity of pain in the postoperative period.

Use of Pain Scale VAS Pain Scale Score: The primary end point is the clinical report of pain. Pain intensity will be assessed using a 100 mm VAS with anchors of "no pain" and "worst pain imaginable" and a 4-point category scale ("none", "mild", "moderate", and "severe") once pre-operatively and over the post-operative observation period at 30-minute intervals during the post- surgical time. The category scale is included for purposes of obtaining a patient-reported assignment of moderate pain (definition of clinically significant pain), and for computing the cut-offs for pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be at least 18 years old.
* Subjects for whom a decision has been made to extract at least two third molars classified as full or partially bony impacted in the mandible and/or maxilla in an outpatient setting under ambulatory general anesthesia.

  1. Full bony: The entire tooth is below the level of the alveolar bone.
  2. Partial bony: A portion of the height of the contour of the tooth is below the level of the alveolar bone.
* Subjects must be physically able to tolerate conventional surgical procedures (ASA I/II)
* Subjects must agree to follow the study protocol.

Exclusion Criteria:

* Subjects who are known to be pregnant or think they may be pregnant. (Female patients will be asked to perform a pregnancy test on the day of surgery to confirm they meet study criteria)
* Subjects with known allergy and/or contradiction to ibuprofen and acetaminophen.
* Subjects with history of alcohol or drug abuse (self-reported).
* Subjects who are currently receiving any anti-inflammatory or pain medication or they suffer from a chronic pain condition.
* Subjects that refuse to participate in the follow up protocol including completing pain diaries.
* Actively infected third molars with swelling, trismus, and/or purulent discharge.
* Subjects for whom the lidocaine with epinephrine is contraindicated (e.g., allergy to drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of IV ibuprofen for post-op pain. | 7 days post-operative
  To determine the efficacy of a single dose of intravenous ibuprofen administered over 5-10 minutes for the preemptive treatment of postoperative pain following third molar extraction.The post operative pain intensity will be measured using (Visual Analog Scale, VAS). A total of 9 pain ratings will be obtained:
  1. Prior to surgery
  2. Immediately after the subject wakes from anesthesia
  3. First onset of pain (typically 45 minutes-1.5 hours after procedure)
  4. 4 hours post-operative
  5. 24 hours post-operative
  6. 48 hours post-operative
  7. 72 hours post-operative
  8. Day 7 post-operative

SECONDARY OUTCOMES:
Pain medication consumption | Post 3rd molar extraction
  To determine any difference in the percentage of pain medications consumed post operatively in both the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Archana Viswanath, BDS,MS, Principal Investigator — Tufts University School of Dental Medicine
Locations (2):
- United States (2):
  - Tufts University School of Dental Medicine Department of Oral and Maxillofacial Surgery, Boston, Massachusetts
  - Tufts University School of Dental Medicine, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hargreaves KM, Troullos ES, Dionne RA. Pharmacologic rationale for the treatment of acute pain. Dent Clin North Am. 1987 Oct;31(4):675-94. PMID 3319716
- [Background] Dionne RA, Khan AA, Gordon SM. Analgesia and COX-2 inhibition. Clin Exp Rheumatol. 2001 Nov-Dec;19(6 Suppl 25):S63-70. PMID 11695255
- [Background] Gordon SM, Brahim JS, Rowan J, Kent A, Dionne RA. Peripheral prostanoid levels and nonsteroidal anti-inflammatory drug analgesia: replicate clinical trials in a tissue injury model. Clin Pharmacol Ther. 2002 Aug;72(2):175-83. doi: 10.1067/mcp.2002.126501. PMID 12189364
- [Background] Ridgway D. Analgesics for acute pain: Meeting the United States Food and Drug Administration's requirements for proof of efficacy. Clin J Pain. 2004 May-Jun;20(3):123-32. doi: 10.1097/00002508-200405000-00001. PMID 15100587
- [Background] Southworth S, Peters J, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen 400 and 800 mg every 6 hours in the management of postoperative pain. Clin Ther. 2009 Sep;31(9):1922-35. doi: 10.1016/j.clinthera.2009.08.026. PMID 19843482
- [Background] Arici S, Gurbet A, Turker G, Yavascaoglu B, Sahin S. Preemptive analgesic effects of intravenous paracetamol in total abdominal hysterectomy. Agri. 2009 Apr;21(2):54-61. PMID 19562533
- [Background] Borisov, D Preemptive analgesia with paracetamol in postoperative analgesia for abdominal surgery: 14AP5-2 European Journal of Anaesthesiology: June 2007 - Volume 24 - Issue - p 179